CLINICAL TRIAL: NCT04077047
Title: Understanding and Developing a Network-based Social Support Intervention to Improve Retention in Human Immunodeficiency Virus (HIV) Care and Antiretroviral Therapy Adherence for Adolescents Living With HIV
Brief Title: Adolescents Living With HIV (ALWH): Social Networks, Adherence and Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00099951; 5K08MH118965-02 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-09-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS
Keywords: Adolescents
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iEngage (Experimental): The intervention is a network-based, social support intervention to improve ALWH retention in HIV care and ART adherence. The specific intervention will be developed during Aim 2 of the study and uses qualitative findings, along with data from Aim 1, to develop an interventions that integrates participant feedback and borrows components from two existing interventions
  Interventions: Behavioral: iEngage

INTERVENTIONS:
Behavioral: iEngage — The intervention is a network-based, social support intervention to improve Adolescents living with HIV (ALWH) retention in HIV care and antiretroviral therapy (ART) adherence
  Other Names: network-based, social support intervention

SUMMARY:
human immunodeficiency virus / acquired immunodeficiency syndrome (HIV/AIDS) is the second leading cause of death in Africa. Adolescents living with HIV (ALWH) are at increased risk for HIV-related morbidity and mortality due to poor retention in HIV care and suboptimal antiretroviral therapy (ART) adherence. Despite having the world's largest population of Adolescents living with HIV (ALWH) (15-24 years, n=870,000), only 14% of South African ALWH are on ART, 12% are retained in HIV care 1-2 years after ART initiation, and 10% are virally suppressed. During treatment interruption, the effects of ART quickly reverse, increasing transmission risk, treatment resistance, and potentially fatal complications. Unless their treatment retention and adherence improves, ALWH will continue to transmit the virus to their sexual partners and die prematurely.

While social support is often viewed as a bridge that joins ALWH to key resources within their environments, little is known about which types of social support are most impactful and from whom within their network, particularly among ALWH in endemic countries. Moreover, many South African ALWH lack social support from key social network members due to lack of HIV status disclosure, increasing their risk for poorer HIV-related outcomes when compare to their disclosed peers. Social network interventions (i.e., those that leverage the resources within one's network to improve behaviors and outcomes) that meet the needs of both ALWH who are disclosed and non-disclosed are needed, but lacking. Such inventions have the potential to facilitate appraisal support, during which ALWH receive targeted assistance with identifying appropriate and trustworthy people in their lives. More broadly, there exists a lack empirically supported interventions aimed at improving retention in HIV care and ART adherence for ALWH in low-middle income countries.

This proposal follows the multiphase optimization strategy (MOST), a comprehensive framework for optimizing and evaluating multicomponent behavioral interventions.

DETAILED DESCRIPTION:
This K08 focuses on the preparation phase, which consists of compiling information from various sources, including behavioral theory, scientific literature, secondary analyses of existing data, and formative research to inform a theoretical model. This model guides intervention-related decisions, such as the selection of intervention components. Piloting of intervention components and the identification and operationalization of an optimization criterion also occur in this phase. The investigators will first use social network analyses to elucidate network characteristics that influence ALWHs' retention and adherence (Aim 1), then use participatory methods to inform intervention development (Aim 2), and lastly assess intervention acceptability, feasibility, safety and evidence of efficacy (Aim 3). Aim 3 is the clinical trial component and described in detail below. Aim 1 will determine how ALWHs' social networks influence their retention in HIV care and ART adherence and Aim 2 will then focus on the development of a network-based, social support intervention to improve ALWH retention in HIV care and ART adherence informed by Aim 1 and other relevant information.

The goal of aim 3 is to assess intervention acceptability, feasibility, safety and evidence of efficacy through open piloting. The investigators will assess intervention acceptability, feasibility, safety, and evidence of efficacy using an iterative process enabling feedback and continuing quality improvement over the course of implementation. This approach involves the piloting of the network intervention developed in Aim 2. The rationale is that the best interventions for ALWH will consider their unique needs and include tailored components. The outcome of this Aim will be a feasible and acceptable social network intervention that will be tested in an adaptive intervention using future grant funding. The hypothesis for aim 3 is that the intervention will be acceptable, feasible, and safe, with trends towards improved ALWH retention in HIV care and ART adherence.

ELIGIBILITY:
Inclusion Criteria:

* reside in study area
* able to provide consent or assent
* agreeable to allowing the research team to have access to their clinic data to assess retention in human immunodeficiency virus- (HIV) care and antiretroviral therapy (ART) adherence
* each Adolescents living with HIV (ALWH) must recruit at least one social network member to participate in the intervention with them

Exclusion Criteria:

* None

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: exit interviews | 12 month follow up
  Measured using exit interviews
Acceptability: exit interviews | 12 month follow up
  Measured using exit interviews

SECONDARY OUTCOMES:
Change in HIV stigma & discrimination | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in HIV knowledge | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in autonomy | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in sense of community | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in basic psychological needs | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in social support | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in trust | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in relationship equity | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in agency | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in future orientation | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in mental health | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in healthcare access | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in physical health | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in housing stability | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in economic support | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in income | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in food security | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in food transportation | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in viral load | baseline, 6 month, and 12 month follow up
  Gathered from existing medical records
Change in ART adherence | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview
Change in retention in HIV care | baseline, 6 month, and 12 month follow up
  may include de novo questionnaire, interview

CONTACTS AND LOCATIONS:
Overall Officials: Tiarney Ritchwood, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States
- Desmond Tutu Health Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT04077047/ICF_000.pdf